CLINICAL TRIAL: NCT02013375
Title: SCD-Haplo: A Phase II Study of HLA-Haploidentical Stem Cell Transplantation to Treat Clinically Aggressive Sickle Cell Disease
Brief Title: SCD-Haplo: Phase II Study of HLA-Haploidentical SCT for Aggressive SCD
Acronym: SCD-Haplo
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Damiano Rondelli, MD (Other)
Responsible Party: Sponsor-Investigator, Damiano Rondelli, MD, Chief, Division of Hematology & Oncology, University of Illinois at Chicago
Organization: University of Illinois at Chicago (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0849
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Alemtuzumab; Whole-Body Irradiation; Cyclophosphamide; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Haploidentical Transplant (Experimental): All subjects will undergo pre-conditioning treatment with alemtuzumab (0.3 mg/kg Day -5, Day -4, Day -3) and total body irradiation (300cGy), followed by stem cell transplant, and post-transplant treatment with cyclophosphamide (50mg/kg/day) and sirolimus (target trough level of 10-15ng/mL).
  Interventions: Procedure: Haploidentical Transplant; Drug: Alemtuzumab; Radiation: Total Body Irradiation; Drug: Cyclophosphamide; Drug: Sirolimus

INTERVENTIONS:
Procedure: Haploidentical Transplant — All subjects will undergo pre-conditioning treatment with alemtuzumab (0.3 mg/kg Day -5, Day -4, Day -3) and total body irradiation (300cGy), followed by stem cell transplant, and post-transplant treatment with cyclophosphamide (50mg/kg/day) and sirolimus (target trough level of 10-15ng/mL).
  Other Names: Mismatched allogeneic bone marrow transplant
Drug: Alemtuzumab — On Day -7, the first test dose of alemtuzumab (0.03 mg/kg) will be administered and on Day -6, the second test dose of alemtuzumab (0.1 mg/kg) will be administered. Alemtuzumab (0.3 mg/kg) will be infused daily on Day -5, -4, and -3.
  Other Names: Campath®
Radiation: Total Body Irradiation — A 300cGy dose of TBI will be administered in a single fraction on Day -2.
Drug: Cyclophosphamide — Cyclophosphamide (50 mg/kg IBW) IV, over approximately 1-2 hours, is given on Day 3 post-transplantation (ideally between 60 and 72 hours after marrow infusion) and on Day 4 (approximately 24 hours after Day 3 cyclophosphamide).
  Other Names: Cytoxan®
Drug: Sirolimus — Sirolimus will be started on Day +5 (at least 24 hours after the completion of the cyclophosphamide infusion). The starting dose will be 12mg followed by 4mg PO daily. Doses will be adjusted to achieve a whole blood trough level of 4 - 12ng/mL.
  Other Names: Rapamune®

SUMMARY:
Related donor stem cell transplantation using the alemtuzumab/ TBI platform has been shown to be a safe strategy to cure severe sickle cell disease. However, due to a lack of suitable donors, many patients cannot benefit from this strategy. Alternative donor sources are desperately needed to fill this gap. Nearly all patients will have a haploidentical family member who would be able to donate. The use of post transplantation cyclophosphamide has greatly improved the outcome of haploidentical stem cell transplantation. The investigators propose to combine this with alemtuzumab/TBI conditioning.

DETAILED DESCRIPTION:
Sickle cell anemia is an inherited form of anemia, a condition in which there aren't enough healthy red blood cells to carry adequate oxygen throughout the body. These patients are at increased risk of death, stroke, frequent pain crises, acute chest syndrome as well as chronic conditions including: lung damage, retinopathy, kidney damage, leg ulcers, and pulmonary hypertension.

There's no cure for most people with sickle cell anemia. However, treatments can relieve pain and help prevent co-morbid conditions associated with sickle cell anemia. Hydroxyurea is the only FDA approved drug to help alleviate symptoms associated with sickle cell disease. The mortality rate is still high in patients using hydroxyurea and a significant percentage of patients still have aggressive disease despite the hydroxyurea treatment. Hydroxyurea therapy also does not seem to prevent the development of many of the complications of sickle cell disease such as pulmonary hypertension.

Historically, stem cell transplantation in sickle cell disease was mainly done in the pediatric population. The options were more limited for adults with sickle cell disease with aggressive disease despite hydroxyurea. Most rely on chronic red blood cell transfusions which carry significant risks of infection, iron overload, and alloimmunization. Alloimmunization refers to the production of antibodies which occurs in up to 50% of patients with sickle cell disease who are on chronic transfusion therapy making further transfusions difficult with a high potential for hemolytic transfusion reactions.

Recently the use of a non-myeloablative stem cell transplantation regimen (relying on immunotherapy instead of chemotherapy) for sickle cell disease in adults showed 88% engraftment rates (30 out of 34 patients) with no GVHD and 0% mortality. However, these transplants used only fully HLA-matched siblings, which are unavailable to all but approximately 14-28% of patients who could benefit from such a transplant at UIC.

A recent study at Johns Hopkins carried out a similar haploidentical (half matched) transplant with 14 sickle cell patients who lacked fully HLA-matched donors. Approximately two years following transplant, 57% of patients successfully engrafted (8 or 14 patients). There were no deaths and only one episode of acute GVHD of the skin which resolved without therapy.

The investigators plan to offer stem cell transplantation to sickle cell patients with aggressive disease who only have a partially matched HLA sibling donor. Haploidentical transplants are considered only for patients with no other standard options available who would normally be treated with supportive (palliative) care or given the option to participate in a clinical trial. Donors who are HLA-haploidentical will be the source of hematopoietic stem cells. Potential donors can include any relative (e.g. parents, offspring, siblings, cousins, aunts/uncles, grandparents).

The related donor stem cell transplantation using the alemtuzumab/TBI platform has been shown to be a safe strategy to cure severe sickle cell disease. However, due to a lack of suitable donors, many patients cannot benefit from this strategy. Alternative donor sources are desperately needed to fill this gap. Nearly all patients will have a haploidentical family member who would be able to donate. The use of post transplantation cyclophosphamide has greatly improved the outcome of haploidentical stem cell transplantation. The investigators propose to combine this with alemtuzumab/TBI conditioning.

The investigational component of this study is the combination of the Alemtuzumab (immunotherapy) and Total Body Irradiation conditioning regimen and the HLA Haploidentical Transplant with post-transplant Cyclophosphamide. Investigators plan to study the engraftment rates (transplant success rates) at Day 60 in sickle cell patients undergoing an HLA haploidentical stem cell transplant with post transplant high dose cyclophosphamide.

ELIGIBILITY:
Patient Eligibility:

* Patients with sickle cell disease are eligible if they have any of the following complications:

  * Stroke or central nervous system event lasting longer than 24 hours
  * Frequent vaso-occlusive pain episodes, defined as ≥ 3 per year requiring emergency room, acute care center, or hospital admissions.
  * Recurrent episodes of priapism, defined as ≥ 2 per year requiring emergency room visits
  * Acute chest syndrome with recurrent hospitalizations, defined as ≥ 2 lifetime events
  * Red-cell alloimmunization (≥ 2 antibodies) during long-term transfusion therapy
  * Bilateral proliferative retinopathy with major visual impairment in at least one eye
  * Osteonecrosis of 2 or more joints
  * Sickle cell nephropathy, defined by a GFR < 90mL/min/1.73m2 or the presence of macroalbuminuria (urine albumin > 300 mg/g creatinine)
  * Pulmonary hypertension, defined by a mean pulmonary artery pressure > 25mmHg
* Age 16-60 years
* Karnofsky performance status of 60 or higher
* Adequate cardiac function, defined as left ventricular ejection fraction ≥ 40%
* Adequate pulmonary function, defined as diffusion lung capacity of carbon monoxide ≥ 50% predicted (after adjustment for hemoglobin concentration)
* Estimated GFR ≥ 50mL/min as calculated by the modified MDRD equation
* ALT ≤ 3x upper limit of normal
* HIV-negative
* Patient is pregnant
* Patient is able and willing to sign informed consent
* Patient has an HLA-haploidentical relative

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2014-04-10 (Actual); Primary Completion 2014-05-31 (Actual); Study Completion 2018-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damiano Rondelli, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Cancer Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects are referred by their primary care physicians to the UIC Sickle Cell clinic for specialty care. Subjects are evaluated to see if they are eligible for studies and if they are, the subject is presented with the option of enrolling into a research study or participating in alternative therapies that have also been presented to the subject.
Groups:
- Haploidentical Transplant: All subjects will undergo pre-conditioning treatment with alemtuzumab (0.3 mg/kg) and total body irradiation (300cGy), followed by stem cell transplant, and post-transplant with cyclophosphamide (50mg/kg/day) and sirolimus (target trough level of 10-15ng/mL).
Period: Overall Study
Arm/Group | Haploidentical Transplant
Started | 2
Completed (Both subjects did not engraft) | 0
Not Completed | 2
Not completed — Did not engraft | 1
Not completed — Did not engraft | 1

BASELINE CHARACTERISTICS:
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants] — Date of birth and age at screening visit
  Participants
    <=18 years | 0
    Between 18 and 65 years | 2
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at screening visit
  Years | 38 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Engraftment Rate
Description: To determine the engraftment at Day +60 following HLA-haploidentical hematopoietic stem cell transplant protocol using immunosuppressive agents and low-dose total body irradiation (TBI) for conditioning and post-transplant cyclophosphamide in patients with sickle cell disease.
Time Frame: Up to Day 60 post-transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 2
Participants | 0

2. Secondary Outcome: Acute & Chronic Complications
Description: To assess the frequency of acute and chronic complications of sickle cell disease during and after HLA-haploidentical hematopoietic stem cell transplantation with this protocol. The acute complications include vaso-occlusive pain episodes, acute chest syndrome, stroke, and priapism. The chronic complications include nephropathy, retinopathy, osteonecrosis, pulmonary artery pressures, cardiomyopathy, and chronic lung disease.
Time Frame: Up to one year post-transplant
Population: No subjects engrafted
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall & Disease-Free Survival
Description: To determine the overall and disease-free survival of patients with sickle cell disease receiving HLA-haploidentical hematopoietic stem cell transplantation with this protocol.
Time Frame: Up to one year post-transplant.
Population: No subjects engrafted
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 0

4. Secondary Outcome: Morbidity & Mortality
Description: To determine the incidence of acute and chronic graft-versus-host disease, the incidence of infectious complications, and the transplant related mortality in sickle cell disease patients after HLA-haploidentical hematopoietic stem cell transplantation with this protocol.
Time Frame: Up to one year post-transplant.
Population: 0 subjects engrafted
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Haploidentical Transplant
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes